CLINICAL TRIAL: NCT00481585
Title: The Biology of Claudin 3 in Primary Human Mammary Epithelial Cell Culture
Status: Terminated | Type: Observational
Why Stopped: study team failed to complete timely reviews, study suspended
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: 07.01.041
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Breast Cancer
Keywords: claudin; electrophysiology; breast; screening
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of the present study is to determine whether or not primary human mammary epithelial cells are competent for use in molecular studies of transepithelial electrophysiology focusing on the function of the tight junction protein claudin 3.

Human breast Tissue will be removed from mastectomy specimens and used as a source to generate epithelial cells for study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of this pilot study are limited to those female patients who are undergoing therapeutic or prophylactic mastectomy procedures conducted by the department of Surgery at HUMC.

Exclusion Criteria:

* From within this population, no exclusion criteria shall be applied based on age, race, ethnicity, gender, HIV status, or menopause.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 13 subjects - Subjects of this pilot study are limited to those female patients who are undergoing therapeutic or prophylactic mastectomy procedures conducted by the department of Surgery at HUMC.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2007-05; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Cell line data study | one year

CONTACTS AND LOCATIONS:
Overall Officials: Erik F Young, Ph.D., Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack Univeristy Medical Center, Hackensack, New Jersey, United States